CLINICAL TRIAL: NCT03943589
Title: An Open-label, Single Arm, Multi-centre, Phase II Study Investigating Safety, Tolerability, Efficacy, Pharmacodynamics and Pharmacokinetics of Imlifidase in Patients With Guillain-Barré Syndrome, in Comparison With Matched Control Patients
Brief Title: A Study of Imlifidase in Patients With Guillain-Barré Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-HMedIdeS-09
Record Dates: First submitted 2019-04-30; First posted 2019-05-09 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Guillain-Barré Syndrome (GBS)
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Mac-1-like protein, Streptococcus

STUDY DESIGN:
Intervention Model Description: Data from patients enrolled in this trial will, if feasible, be compared with an external control group consisting of patients from the IGOS database (International Guillain-Barré Syndrome Outcome Study, ClinicalTrials.gov Identifier: NCT01582763).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imlifidase (Experimental): One (1) dose of imlifidase, 0.25 mg/kg, will be administered IV over 30 minutes, Day 1.
  IVIg, 0.4 g/kg, will be administered for 5 consecutive Days, starting on Day 3 at least 48 h after imlifidase administration.
  Interventions: Drug: Imlifidase

INTERVENTIONS:
Drug: Imlifidase — All subjects will receive imlifidase (Day 1) prior to standard care IVIg
  Other Names: Hansa Medical-Immunoglobulin G degrading enzyme of Streptococcus pyogenes (HMED-IdeS), IdeS, IgG endopeptidase

SUMMARY:
The study participants are patients which have been diagnosed with Guillain-Barré Syndrome (GBS) and are planned to receive treatment with intravenous immunoglobulin (IVIg). IVIg is a standard of care treatment for GBS patients. The patients in this study will be treated with the study medicine imlifidase on day 1, and with IVIg on days 3-7.

The purpose of this study is to investigate the safety and effectiveness of imlifidase in patients diagnosed with GBS.

DETAILED DESCRIPTION:
This is an open-label, single arm, multi-centre, phase II study of imlifidase in combination with standard care IVIg in patients with GBS.

The study will recruit approximately 30 patients who are eligible for IVIg treatment based on current practice (i.e. GBS disability score >3 and within 10 days of onset of weakness). All patients will receive imlifidase (Day 1) prior to standard care IVIg.

There is growing body of evidence suggesting that GBS is an antibody-mediated disorder. In addition to supportive care, IVIg and Plasma Exchange (PE) are the two main immunological treatment options aimed at attenuating the autoreactive humoral immune response. Imlifidase is an IgG degrading enzyme with strict specificity. The hypothesis is that reduction of pathological antibodies may result in aborted progression, quicker recovery and less severe disease.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent obtained before any study-related procedures.
2. Willingness and ability to comply with the protocol.
3. Male or female aged ≥18 years at the time of screening.
4. GBS diagnosed according to National Institute of Neurological Disorders and Stroke (NINDS) diagnostic criteria (Asbury et al. 1990).
5. Onset of weakness due to GBS is not more than 10 days prior to screening.
6. Unable to walk unaided for >10 meters (grade ≥ 3 on GBS DS).
7. IVIg treatment being considered.
8. Women of child-bearing potential willing or able to use at least one highly effective contraceptive method from the day of treatment until at least 6 months after the dose of imlifidase if not abstinent. In the context of this study, an effective method is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
9. Men willing to use double-barrier contraception from the day of treatment until at least 2 months after the dose of imlifidase if not abstinent.

Exclusion Criteria:

1. Previous treatment with imlifidase.
2. Previous IVIg treatment within 28 days prior to imlifidase treatment.
3. Subjects who are being considered for, or already on, PE.
4. Women of child-bearing potential willing or able to use at least one highly effective contraceptive method from the screening visit until at least 180 days following imlifidase dosing.
5. Breastfeeding or pregnancy
6. Clinical evidence of a polyneuropathy of another cause e.g. diabetes mellitus (except mild sensory), alcoholism, vitamin deficiency, or porphyria.
7. Known selective immunoglobulin A (IgA) deficiency.
8. Hypersensitivity to IVIg or to any of the excipients.
9. Immunosuppressive treatment (e.g. azathioprine, cyclosporine, mycophenolate mofetil, tacrolimus, sirolimus or > 20 mg prednisolone daily) during the last month.
10. Subject known to have a severe concurrent disease, e.g. malignancy, severe cardiovascular disease and severe chronic obstructive pulmonary disease (COPD).
11. Any condition that in the opinion of the investigator could increase the subject's risk by participating in the study or confound the outcome of the study.
12. Known mental incapacity or language barriers precluding adequate understanding of the Informed Consent information and the study activities.
13. Subjects with clinical signs of ongoing infection.
14. Subjects should not have received other investigational drugs within 5 half-lives prior to imlifidase dosing.
15. Present or history of thrombotic thrombocytopenic purpura (TTP), or known familial history of TTP.
16. Positive PCR test for SARS-CoV-2 virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Chair — Hansa Biopharma AB
Locations (11):
- France (7):
  - CHU Le Kremlin-Bicêtre. Service Neurologie, Le Kremlin-Bicêtre, Paris
  - CHU Bordeaux - Hôpital Pellegrin Tripode, Bordeaux
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Hôpital de la Timone - Centre de référence des maladies neuromusculaires et de la SLA, Marseille
  - CHU de Montpellier, Hôpital Gui de Chauliac, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Service de neurologie, Hôpitaux Universitaires de Strasbourg, Strasbourg
- Netherlands (2):
  - Amsterdam UMC, Amsterdam
  - Erasmus Medical Centre, Rotterdam
- United Kingdom (2):
  - Queen Elizabeth University Hospital Glasgow, Glasgow
  - Oxford University Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Imlifidase: One (1) dose of imlifidase, 0.25 mg/kg, will be administered IV over 30 minutes, Day 1.
  IVIg, 0.4 g/kg, will be administered for 5 consecutive Days, starting on Day 3 at least 48 h after imlifidase administration.
  Imlifidase: All subjects will receive imlifidase (Day 1) prior to standard care IVIg
Period: Overall Study
Arm/Group | Imlifidase
Started | 30
Completed | 28
Not Completed | 2
Not completed — Death | 1
Not completed — Diagnosed with encephalomyelitis | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24
  Asian | 2
  Black or African American | 1
  Other | 3
Region of Enrollment [Number; unit: participants]
  Netherlands | 1
  United Kingdom | 3
  France | 26
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.8 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Guillain Barré Syndrome Disability Score (GBS DS) - Time to Improve by at Least 1 Grade
Description: Efficacy is assessed as proportion of subjects with improvement of one (1) or more grades in disability outcome on the 6-point GBS DS over time.
  The 6-point Guillain Barré Syndrome disability score (GBS DS) is a widely accepted and easily obtainable scoring system used to assess disability status of GBS subjects. The DS score is as follows: 0=Healthy, 1=Minor symptoms and capable of running (subjects must be asked to run), 2=Able to walk independently 10 meters or more but unable to run, 3=Able to walk more than 10 meters across an open space with help, 4=Bedridden or chair bound, 5=Needing mechanical ventilation, 6=Dead
Time Frame: Baseline to Day 360
Population: The full analysis set (FAS) consists of data from all dosed patients having a confirmed GBS diagnosis, i.e., patients re-evaluated and having change in diagnosis (incorrectly diagnosed with GBS at trial entry) were excluded.
Measure: Median (Full Range); unit: days
Arm/Group | Imlifidase
Number analyzed (Participants) | 27
days | 6.0 [3.0 to 16.0]

2. Primary Outcome: Guillain Barré Syndrome Disability Score (GBS DS) - Time to Improve by at Least 2 Grades
Description: as for outcome 1
Time Frame: Baseline to Day 360
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Imlifidase
Number analyzed (Participants) | 27
days | 16.0 [8.0 to 92.0]

3. Primary Outcome: Guillain Barré Syndrome Disability Score (GBS DS) - Ability to Walk Unaided
Description: Efficacy is assessed as proportion of subjects able to walk unaided (i.e. GBS DS=2) over time
Time Frame: Baseline to Day 360
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 27
Participants
  Baseline | 0
  Day 2 | 4
  Day 3 | 5
  Day 4 | 9
  Day 5 | 9
  Day 6 | 9
  Day 7 | 10
  Day 8 | 10
  Day 15 | 13
  Day 29 | 14
  Day 57 | 18
  Day 92 | 20
  Day 180 | 23
  Day 360 | 24

4. Primary Outcome: Proportion of Patients Who Are Able to Run Over Time (GBS DS≤1)
Description: Efficacy is assessed as proportion of patients able to run (i.e. Guillain Barré Syndrome disability score [GBS DS] ≤1) over time
Time Frame: Baseline to Day 360
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 27
Participants
  Baseline | 0
  Day 2 | 0
  Day 3 | 0
  Day 4 | 0
  Day 5 | 1
  Day 6 | 1
  Day 7 | 2
  Day 8 | 4
  Day 15 | 5
  Day 29 | 9
  Day 57 | 11
  Day 92 | 15
  Day 180 | 17
  Day 360 | 18

5. Primary Outcome: Mean MRC Sum Score Over Time
Description: Efficacy is assessed as Medical Research Council (MRC) sum score over time.
  The MRC sum score is widely used to assess the motor impairment in subjects with peripheral neuropathies. It is a sum score of power in 6 muscle groups on each side (abduction of arm, flexion of forearm, extension of the wrist, hip flexion, and extension of knee and dorsal flexion of the foot). The sum of these scores ranges from 0 (total paralysis) to 60 (normal power). It provides valuable information about the muscle strength. Change in MRC sum score helps in identification of GBS patients with treatment related fluctuation or exacerbation. The individual MRC grades are defined as follows: 0=No visible contraction,1=Visible contraction without movement of the limb, 2=Movement of the limb but not against gravity, 3=Movement against gravity (almost full range), 4=Movement against gravity and resistance, 5=Normal
Time Frame: Baseline until Day 180
Population: The full analysis set (FAS) consists of data from all dosed patients having a confirmed GBS diagnosis, i.e., patients re-evaluated and having change in diagnosis (incorrectly diagnosed with GBS at trial entry) were excluded.
  26 patients with data at Day 6 and Day 8, 25 patients with data at Day 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imlifidase
Number analyzed (Participants) | 27
score on a scale
  Baseline | 39.1 (13.88)
  Day 2 | 42.0 (14.66)
  Day 4 | 47.5 (14.58)
  Day 6: number analyzed (Participants) | 26
  Day 6 | 49.7 (13.70)
  Day 8: number analyzed (Participants) | 26
  Day 8 | 50.0 (13.80)
  Day 15: number analyzed (Participants) | 25
  Day 15 | 51.8 (12.09)
  Day 29 | 49.1 (17.41)
  Day 57 | 49.0 (18.39)
  Day 92 | 51.8 (16.22)
  Day 180 | 54.1 (12.40)

6. Primary Outcome: Change From Baseline in MRC Sum Score Over Time
Description: Efficacy is assessed as change in Medical Research Council (MRC) sum score.
  The MRC sum score is widely used to assess the motor impairment in subjects with peripheral neuropathies. It is a sum score of power in 6 muscle groups on each side (abduction of arm, flexion of forearm, extension of the wrist, hip flexion, and extension of knee and dorsal flexion of the foot). The sum of these scores ranges from 0 (total paralysis) to 60 (normal power). It provides valuable information about the muscle strength. Change in MRC sum score helps in identification of GBS patients with treatment related fluctuation or exacerbation. The individual MRC grades are defined as follows: 0=No visible contraction,1=Visible contraction without movement of the limb, 2=Movement of the limb but not against gravity, 3=Movement against gravity (almost full range), 4=Movement against gravity and resistance, 5=Normal
Time Frame: Baseline until Day 180
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imlifidase
Number analyzed (Participants) | 27
score on a scale
  Day 2 | 2.9 (8.23)
  Day 4 | 8.4 (9.19)
  Day 6: number analyzed (Participants) | 26
  Day 6 | 10.3 (9.81)
  Day 8: number analyzed (Participants) | 26
  Day 8 | 10.7 (10.21)
  Day 15: number analyzed (Participants) | 25
  Day 15 | 11.2 (10.42)
  Day 29 | 10.0 (12.99)
  Day 57 | 9.9 (14.59)
  Day 92 | 12.7 (12.96)
  Day 180 | 15.0 (10.62)

7. Primary Outcome: Mean R-ODS Over Time
Description: The patients have rated their ability to perform different common activities using the Rasch-built overall disability score (R-ODS) questionnaire.
  R-ODS is a linearly weighted disease specific scale, which captures activities and social participation limitation in patients with immune-mediated neuropathies, including GBS. The questionnaire comprises 24 items ranging from ability to read a book or newspaper (as the easiest item to accomplish) to ability to run (most difficult item to accomplish). The response options for each item are: 0=Not possible, 1=Possible with effort, 2=Easy to perform. The obtained raw summed score is subsequently translated to a centile metric ranging from 0 (most severe disability) to 100 (no disability at all).
Time Frame: Baseline to Day 360
Population: The full analysis set (FAS) consists of data from all dosed patients having a confirmed GBS diagnosis, i.e., patients re-evaluated and having change in diagnosis (incorrectly diagnosed with GBS at trial entry) were excluded.
  24 patients with data at Day 15, 26 patients with data at Day 8, Day 57, Day 92 and day 360.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imlifidase
Number analyzed (Participants) | 27
score on a scale
  Baseline | 23.7 (15.26)
  Day 8: number analyzed (Participants) | 26
  Day 8 | 41.9 (28.01)
  Day 15: number analyzed (Participants) | 24
  Day 15 | 46.2 (26.87)
  Day 29 | 52.6 (33.12)
  Day 57: number analyzed (Participants) | 26
  Day 57 | 57.2 (34.54)
  Day 92: number analyzed (Participants) | 26
  Day 92 | 63.5 (32.50)
  Day 180 | 70.0 (29.17)
  Day 360: number analyzed (Participants) | 26
  Day 360 | 73.8 (24.36)

8. Primary Outcome: Change From Baseline in R-ODS Over Time
Description: as for outcome 7
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imlifidase
Number analyzed (Participants) | 27
score on a scale
  Day 8: number analyzed (Participants) | 26
  Day 8 | 17.2 (22.3)
  Day 15: number analyzed (Participants) | 24
  Day 15 | 20.8 (21.4)
  Day 29 | 28.8 (25.3)
  Day 57: number analyzed (Participants) | 26
  Day 57 | 34.5 (26.5)
  Day 92: number analyzed (Participants) | 26
  Day 92 | 40.8 (24.6)
  Day 180 | 46.3 (22.7)
  Day 360: number analyzed (Participants) | 26
  Day 360 | 50.5 (19.3)

9. Primary Outcome: Days in Hospital
Description: The number of days the patients were admitted to hospital
Time Frame: Baseline to Day 360
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
days | 32.5 (43.5)

10. Primary Outcome: Time in an ICU
Description: Efficacy is assessed as time in an intensive care unit (ICU)
Time Frame: Baseline until Day 360
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
Participants
  Admitted 0 days | 18
  Admitted 2-11 days | 9
  Admitted 106-113 days | 2
  Admitted 172 days | 1

11. Primary Outcome: Need for Mechanical Ventilation
Time Frame: Baseline until Day 180
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
Participants
  Screening | 0
  Day 1 to Day 90 | 1
  Day 5 to Day 102 | 1
  Day 9 to Day 90 and Day 103 to Day 180 | 1

12. Primary Outcome: Patient's Health State Over Time as Assessed by EQ VAS
Description: Quality of Life will be assessed using the EurQol group's EurQol - 5 dimension (EQ-5D) Health questionnaire.
  The EQ-5D consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ VAS records the patient's self-rated health on a vertical scale, where score 100 is 'The best health you can imagine' and score 0 is the 'The worst health you can imagine'.
Time Frame: Day 8, Day 15, Day 29, Day 57, Day 92, Day 180, and Day 360
Population: Safety analysis set 27 patients with data at Day 92 and Day180, 26 patients with data at Day 8 and Day 360, 25 patients with data at Day 29 and Day 57, 24 patients with data at Day 15.
Measure: Mean (Standard Deviation); unit: EQ-5D-5L VAS score
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
EQ-5D-5L VAS score
  Day 8: number analyzed (Participants) | 26
  Day 8 | 49.7 (23.7)
  Day 15: number analyzed (Participants) | 24
  Day 15 | 61.3 (24.8)
  Day 29: number analyzed (Participants) | 25
  Day 29 | 67.3 (21.0)
  Day 57: number analyzed (Participants) | 25
  Day 57 | 68.8 (25.1)
  Day 92: number analyzed (Participants) | 27
  Day 92 | 75.2 (23.9)
  Day 180: number analyzed (Participants) | 27
  Day 180 | 78.6 (20.6)
  Day 360: number analyzed (Participants) | 26
  Day 360 | 79.4 (18.6)

13. Secondary Outcome: PK Profile of Imlifidase: Cmax
Description: Cmax=Maximum observed plasma concentration of imlifidase following dosing
Time Frame: Within 2 hours before imlifidase dose until Day 15
Population: Sampling for PK evaluation was performed for the first 16 patients included in the trial
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Imlifidase
Number analyzed (Participants) | 16
µg/mL | 5.5 (17.0)

14. Secondary Outcome: PK Profile of Imlifidase: Tmax
Description: Tmax=Time point for maximum observed plasma concentration of imlifidase following dosing
Time Frame: Within 2 hours before imlifidase dose until Day 15
Population: Sampling for PK evaluation was performed for the first 16 patients included in the trial.
Measure: Median (Full Range); unit: hours
Arm/Group | Imlifidase
Number analyzed (Participants) | 16
hours | 0.74 [0.47 to 2.07]

15. Secondary Outcome: PK Profile of Imlifidase: AUC
Description: AUC=Area under the imlifidase plasma concentration versus time curve
Time Frame: Within 2 hours before imlifidase dose until Day 15
Population: Sampling for PK evaluation was performed for the first 16 patients included in the trial. The time-concentration profile of imlifidase has previously been shown to generally fit a 2-compartment model. 9 out of the 16 patients could be fitted with a 2-compartment model.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h×µg/mL
Arm/Group | Imlifidase
Number analyzed (Participants) | 9
h×µg/mL | 45.0 (54.9)

16. Secondary Outcome: PK Profile of Imlifidase: t1/2
Description: t1/2=Terminal half-life of imlifidase
Time Frame: Within 2 hours before imlifidase dose until Day 15
Population: Sampling for PK evaluation was performed for the first 16 patients included in the trial. The time-concentration profile of imlifidase has previously been shown to generally fit a 2-compartment model. 9 out of the 16 patients could be fitted with a 2-compartment model.
  Please note, harmonic mean is used for the t½ α and t½ β.
Measure: Mean (Full Range); unit: hours
Arm/Group | Imlifidase
Number analyzed (Participants) | 9
hours
  t½ initial phase (α) | 1.73 [0.95 to 3.26]
  t½ terminal phase (β) | 30.58 [9.13 to 92.79]

17. Secondary Outcome: PK Profile of Imlifidase: CL
Description: CL=Clearance of imlifidase
Time Frame: Within 2 hours before imlifidase dose until Day 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | Imlifidase
Number analyzed (Participants) | 9
mL/h/kg | 5.6 (54.9)

18. Secondary Outcome: PK Profile of Imlifidase: V
Description: V=Volume of distribution
Time Frame: Within 2 hours before imlifidase dose until Day 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | Imlifidase
Number analyzed (Participants) | 9
L/kg
  Volume of distribution at steady state (Vss) | 0.2 (41.1)
  Volume of distribution during the elimination phase (Vz) | 0.3 (40.7)

19. Secondary Outcome: Pharmacodynamics - IgG Level in Serum Over Time
Description: The pharmacodynamic (PD) effect of imlifidase is assessed as the elimination of IgG. IgG is cleaved by imlifidase in two steps, the first cut generates single-cleaved IgG (scIgG), and the second cut generates one F(ab')2 fragment and one Fc fragment. The IgG concentration measured in serum using the MSD technology is the sum of intact IgG and scIgG and a decrease in the measured IgG concentration therefore represents complete cleavage of the IgG molecule to Fc and F(ab')2 fragments. For the first 16 patients included in the trial a more frequent PD sampling schedule was conducted. After amending the protocol a less frequent PD sampling schedule was applied.
Time Frame: Within 2 hours before imlifidase dose until Day 15
Population: 16 patients analyzed at Day 4, Day 5, Day 6 and Day 7 as the protocol was amended after 16 patients were included and a less frequent PD sampling schedule was applied.
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
mg/mL
  Day 1, pre-dose | 10.8 (4.5)
  Day 2, 24 hours after dose | 1.3 (3.5)
  Day 3, before IVIg administration | 1.6 (3.5)
  Day 4, before IVIg administration: number analyzed (Participants) | 16
  Day 4, before IVIg administration | 8.6 (2.3)
  Day 5, before IVIg administration: number analyzed (Participants) | 16
  Day 5, before IVIg administration | 14.3 (1.9)
  Day 6, before IVIg administration: number analyzed (Participants) | 16
  Day 6, before IVIg administration | 18.1 (4.0)
  Day 7, before IVIg administration: number analyzed (Participants) | 16
  Day 7, before IVIg administration | 20.8 (5.5)
  Day 8 | 28.6 (9.2)
  Day 15 | 22.5 (10.0)

20. Secondary Outcome: Immunogenicity - Anti-imlifidase Antibodies (ADA) Over Time
Description: Anti-imlifidase IgG antibodies (ADA) in serum.
Time Frame: Within 2 hours before imlifidase dose until Day 180
Population: 28 patients have data at Day 29, Day 57, Day 92, and Day 180
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Imlifidase
Number analyzed (Participants) | 30
mg/L
  Day 1, pre-dose | 11.1 (17.1)
  Day 2, 24 hours after dose | 4.0 (9.6)
  Day 3, before IVIg administration | 4.5 (12.2)
  Day 8 | 474.5 (909.0)
  Day 15 | 2811.9 (3772.6)
  Day 29: number analyzed (Participants) | 28
  Day 29 | 2120.1 (2813.7)
  Day 57: number analyzed (Participants) | 28
  Day 57 | 1060.3 (1086.5)
  Day 92: number analyzed (Participants) | 28
  Day 92 | 722.1 (806.8)
  Day 180: number analyzed (Participants) | 28
  Day 180 | 336.0 (318.9)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for 1 year (i.e., from the timepoint the patient signed the informed consent form (ICF) until Day 360.
Description: AEs were either spontaneously reported, reported in response to an open question, or revealed by observation.
  A treatment-emergent AE (TEAE) is any AE occurring after imlifidase dosing and within 29 days.
  The listed non-serious AEs includes both pre-TEAEs, TEAEs and post-TEAEs. 18 SAEs have been reported, 9 of which were treatment-emergent. All SAEs are listed.
Arm/Group | Imlifidase
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 7/30
Other Adverse Events (participants affected / at risk) | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imlifidase (N=30)
False positive investigation result (Investigations) | 1 (1) — Covid false positive
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 3 (4)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1)
Central nervous system inflammation (Nervous system disorders) | 1 (1)
Demyelination (Nervous system disorders) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imlifidase (N=30)
Constipation (Gastrointestinal disorders) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Corona virus infection (Infections and infestations) | 5 (5)
Pneumonia (Infections and infestations) | 3 (4)
Escherichia urinary tract infection (Infections and infestations) | 3 (3)
Urinary tract infection bacterial (Infections and infestations) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Viral rash (Infections and infestations) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 3 (3)
Facial paralysis (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 2 (2)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Idiopathic intracranial hypertension (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Piriformis syndrome (Nervous system disorders) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
C-reactive protein increased (Investigations) | 3 (4)
Liver function test abnormal (Investigations) | 2 (2)
White blood cell count increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Haemoglobin urine present (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (1)
Staphylococcus test positive (Investigations) | 1 (1)
Troponin I increased (Investigations) | 1 (1)
Urine ketone body present (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 3 (3)
Hallucination (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Intensive care unit delirium (Psychiatric disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (7)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Chills (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Vessel puncture site phlebitis (General disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectas (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1)
Lagophthalmos (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 3 (3)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cutaneous calcification (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the study, one or more manuscripts for joint publication may be prepared in collaboration between the investigator(s) offered authorship and Hansa Biopharma.

Any confidential information relating to imlifidase or the study, including any data and results from the study will be the exclusive property of Hansa Biopharma AB. The investigators and any other persons involved in the trial will protect the confidentiality of the proprietary information belonging to Hansa Biopharma AB

DOCUMENTS (2):
  • Study Protocol (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT03943589/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT03943589/SAP_001.pdf